CLINICAL TRIAL: NCT06943365
Title: Circulating Anti-TREK-1 Autoantibodies as Diagnostic and Prognostic Biomarkers in Short-Coupled Ventricular Fibrillation
Brief Title: Role of Anti-TREK-1 Autoantibodies in SCVF
Acronym: TRACK-VF
Status: Enrolling by invitation | Type: Observational
Sponsor: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Christian Steinberg, MD, Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Other Study IDs: MP-10-2025-4338
Record Dates: First submitted 2025-04-06; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Short-coupled Ventricular Fibrillation; Idiopathic Ventricular Fibrillation
Keywords: SCVF; anti-TREK-1
MeSH Terms: conditions — Paroxysmal ventricular fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SCVF: Probands with diagnosis of SCVF
  Interventions: Other: Repeat plasma screening for the presence or absence of anti-TREK-1 autoantibodies; Genetic: DPP6 risk haplotype

INTERVENTIONS:
Other: Repeat plasma screening for the presence or absence of anti-TREK-1 autoantibodies — Semiquantitative measure of circulating anti-TREK-1 autoantibodies in plasma of study participants using a peptid microarray
Genetic: DPP6 risk haplotype — Systematic genetic screening for the Dutch DPP6 risk haplotype in all study participants and correlation of results with the presence or absence of anti-TREK-1 autoantibodies

SUMMARY:
Short-coupled ventricular fibrillation (SCVF) is a lethal, primary electrical disorder and an important cause of unexplained cardiac arrest.1 Recent work from our group suggests that a substantial proportion of SCVF cases is associated to circulating autoantibodies targeting TREK-1, a cardiac potassium channel, resulting in an abnormal gain-of-function which is the prerequisite for the SCVF phenotype.2 This proposal is a translational multicenter study to validate anti-TREK-1 autoantibodies as a diagnostic and prognostic biomarker in a large, diversified cohort of SCVF patients (Figure 1). Functional, cellular experiments in patient-derived hiPSC cardiomyocytes and Purkinje cells will be performed to explore the cell type-specific role of TREK-1 in arrhythmogenesis, while single-nuclear RNA sequencing (snRNA-seq) will allow us to establish the transcriptomic profile (Figure 1). These results will identify the cellular substrate for SCVF.

DETAILED DESCRIPTION:
Please refer to the uploaded study protocol

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of SCVF as per current criteria
* Willingness to provide written informed consent

Exclusion Criteria:

- SCVF patients < age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort study of SCVF probands
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of anti-TREK-1 autoantibodies at three different time points | 12 months
  Plasma concentrations of anti-TREK-1 autoantibodies (semiquantitative measure using a peptide microarray at three predefined time points

SECONDARY OUTCOMES:
Time-dependent variability of plasma concentrations of anti-TREK-1 autoantibodies | 12 months
  Repeat plasma sampling to assess the presence/absence of anti-TREK-1 autoantibodies and time-dependent variability of antibody expression
Impact of anti-TREK-1 autoantibodies on disease severity | 12 months
  Correlation of the presence (plasma concentration) of anti-TREK-1 autoantibodies with recurrent VF, electrical storm and appropriate ICD therapies

CONTACTS AND LOCATIONS:
Overall Officials: Christian Steinberg, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut universitaire de cardiologie et pneumologie de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steinberg C. Short-Coupled Ventricular Fibrillation. Card Electrophysiol Clin. 2023 Sep;15(3):331-341. doi: 10.1016/j.ccep.2023.05.004. Epub 2023 Jun 18. PMID 37558303
- [Background] Steinberg C, Davies B, Mellor G, Tadros R, Laksman ZW, Roberts JD, Green M, Alqarawi W, Angaran P, Healey J, Sanatani S, Leather R, Seifer C, Fournier A, Duff H, Gardner M, McIntyre C, Hamilton R, Simpson CS, Krahn AD. Short-coupled ventricular fibrillation represents a distinct phenotype among latent causes of unexplained cardiac arrest: a report from the CASPER registry. Eur Heart J. 2021 Jul 31;42(29):2827-2838. doi: 10.1093/eurheartj/ehab275. PMID 34010395
- [Background] Li J, Janin A, Patoughi M, Gaudreault N, Kis L, Moha Ou Maati H, Bosse Y, Steinberg C. Circulating Autoantibodies Targeting TREK-1 in Patients With Short-Coupled Ventricular Fibrillation. Circulation. 2024 Dec 10;150(24):1944-1954. doi: 10.1161/CIRCULATIONAHA.124.070284. Epub 2024 Sep 24. PMID 39315453